CLINICAL TRIAL: NCT02468466
Title: Impact of a Community-based Screening and Educational Intervention for Depression on Suicide Rates Among Japanese Middle-aged Adults
Brief Title: A Community-based Depression Screening Intervention for Middle-aged Suicide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aomori University of Health and Welfare (Other)
Responsible Party: Principal Investigator, Hirofumi Oyama, Faculty of Health Sciences, Aomori University of Health and Welfare
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KAKENHI #70404829
Record Dates: First submitted 2015-06-03; First posted 2015-06-10 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-06

CONDITIONS: Suicide
Keywords: suicide; prevention
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Multi-level suicide prevention programs (Experimental): The study team, including staff members from the intervention municipalities, provided each municipality with a standardized form of the work plan used in our study. The intervention municipality autonomously conducted the intervention program during the implementation period.
  Interventions: Behavioral: Multi-level suicide prevention programs
- Community intervention as usual (Active Comparator): Suicide prevention program as usual
  Interventions: Behavioral: Suicide prevention program as usual

INTERVENTIONS:
Behavioral: Multi-level suicide prevention programs — The intervention included both screening and educational components. The screening component invited residents aged 36-64 years to participate in a two-step screening program. In the initial screening, a self-report questionnaire were mailed to all of those residents in the priority districts with a past high suicide rate. The second stage was conducted for the participants who screened positive though a semi-structural interview. Based on the results, participants who were diagnosed with a major depressive episode were provided with a referral to a psychiatry and support for treatment adherence. Written feedback on the screening results was mailed to all respondents. The educational component was implemented through workshops open to the general public (3 times every year) and local public newsletters (twice every year) designed to improve access and adherence to treatment and to reduce stigma associated with suicide and depression.
  Arms: Multi-level suicide prevention programs
Behavioral: Suicide prevention program as usual — Usual mental health program (not including depression screening among middle-aged)
  Arms: Community intervention as usual

SUMMARY:
The purpose of this study is to examine the effectiveness of a community-based depression-screening program for suicide prevention among middle-aged adults, the investigators conducted a quasi-experimental intervention study, using a parallel cluster design with communities at municipal level as the unit of allocation and individuals as the unit of analysis.

DETAILED DESCRIPTION:
Suicide is a major cause of premature death, particularly among middle-aged adults, in the majority of Western and Asian countries. A strong association of suicide and depression often indicates the necessity of a high-risk approach for suicide prevention. Improvements in identification and treatment can lead to better depression outcomes and suicide prevention. The investigators hypothesize that a 4-year community-based intervention, consisting of universal depression screening and subsequent care support in the target areas and health education programs, would result in reduced suicide rates among the middle-aged adult population in areas with a high suicide rate.

ELIGIBILITY:
Inclusion Criteria:

* A municipal area located in the following 4 Aomori Second Medical Zones: Hachinohe, Kamitosan, Aomori, and Tsugaru.
* A municipal area with the higher suicide rate than the prefectural average.
* A municipal area having the sufficient and coverable size to serve the intervention (population 10,000-99,999).

Exclusion Criteria:

* A municipal area receiving further intervention including a depression screening for middle-aged adults.

Ages: 36 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 89700 (Actual)
Dates: Start 2005-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change in suicide rates among adults aged 40-64 years between the 4-year pre- and implementation periods. | 4 years pre versus 4 years post

SECONDARY OUTCOMES:
Invitation rate in the screening component | 4 years post
Participation rate in the screening component | 4 years post

CONTACTS AND LOCATIONS:
Overall Officials: Hirofumi Oyama, MD, PhD, Study Director — Aomori University of Health and Welfare
Locations (11):
- Japan (11):
  - Control group, Fujisaki, Aomori
  - Intervention group, Gonohe, Aomori
  - Intervention group, Hashikami, Aomori
  - Intervention group, Hirakawa, Aomori
  - Control group, Hiranai, Aomori
  - Intervention group, Nanaku, Aomori
  - Intervention group, Oirase, Aomori
  - Control group, Ōwani, Aomori
  - Control group, Rokunohe, Aomori
  - Control group, Tohoku, Aomori
  - Control group, Towada, Aomori

REFERENCES:
- [Background] Oyama H, Sakashita T. Effects of universal screening for depression among middle-aged adults in a community with a high suicide rate. J Nerv Ment Dis. 2014 Apr;202(4):280-6. doi: 10.1097/NMD.0000000000000119. PMID 24647214
- [Background] Oyama H, Sakashita T. Differences in specific depressive symptoms among community-dwelling middle-aged Japanese adults before and after a universal screening intervention. Soc Psychiatry Psychiatr Epidemiol. 2014 Feb;49(2):251-8. doi: 10.1007/s00127-013-0735-6. Epub 2013 Jul 4. PMID 23824236